CLINICAL TRIAL: NCT00135564
Title: Evaluate the Persistence and Immune Memory Induced by a Primary Vaccination Course With GSK Biologicals' MenC-TT (1 Formulation) & GSK Biologicals' Hib-MenC-TT (2 Formulations) or Meningitec™ in Healthy Toddlers Aged 12-15 Months Primed in Study 711202/001
Brief Title: Study to Evaluate GlaxoSmithKline (GSK) Biologicals' MenC-TT and Hib-MenC-TT or Meningitec™ in Healthy Toddlers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 711202/008
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Meningococcal
Keywords: Haemophilus Influenzae type b/Meningococcal (vaccine); Prophylaxis meningococcal serogroup C disease, Hib diseases
MeSH Terms: conditions — Meningococcal Infections

INTERVENTIONS:
Biological: MenC-TT
Biological: Hib-MenC-TT

SUMMARY:
The purpose of this booster vaccination study is to evaluate the persistence and immune memory induced by a three-dose primary vaccination course with GSK Biologicals' MenC-TT (Neisseria meningitidis group C polysaccharide-tetanus toxoid) and GSK Biologicals' Hib-MenC-TT (Haemophilus influenzae type b-MenC-TT) or Meningitec™ vaccines in healthy toddlers aged 12-15 months by giving them a 1/5th dose of Mencevax™ ACWY.

DETAILED DESCRIPTION:
The study is an extension of the primary vaccination study 711202/001 (MenC-TT-001). It comprises 5 groups: 4 parallel groups of toddlers vaccinated in study 711202/001 (group vaccinated with Meningitec™ is control group 1) and 1 group of naive subjects (no previous vaccination against MenC disease, control group 2). All subjects receive 1/5th dose Mencevax™ ACWY and a concomitant dose of Infanrix hexa®. 2 blood samples: prior to and 1 month after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy toddlers (12-15 m) with at least 1 dose of the 3-dose vaccination course of MenC or Hib-MenC vaccine in study 711202/001, OR without previous vaccination against MenC disease but with completed primary vaccination according to the German Standing Committee on Immunization (STIKO) recommendation at least 6 months before enrolment

Exclusion Criteria:

* Previous/intercurrent booster vaccination against OR history of OR exposure to diphtheria, pertussis, tetanus, polio, hepatitis B, Hib and/or meningococcal disease.
* Planned administration/administration of a vaccine within 30 d preceding study vaccination and until study end with the exception of Infanrix hexa®.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of any neurologic disorders or seizures, of allergic disease/reactions likely to be exacerbated by any component of the vaccines

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2003-01; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Prior to dose 1, 1 month (m) post doses 2, 3: antibody levels to SBA-MenC, anti-polysaccharide C (PSC) in all groups

SECONDARY OUTCOMES:
Prior to dose 1, 1 m post doses 2, 3: anti-PRP
Prior to dose 1, 1 m post dose 3: anti-diphtheria, T, HBs, polio, PT, FHA, PRN
Solicited (days [d] 0-7), unsolicited (up to 30 d) adverse events (AEs) after each dose
Serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Result] Schmitt HJ, Maechler G, Habermehl P, Knuf M, Saenger R, Begg N, Boutriau D. Immunogenicity, reactogenicity, and immune memory after primary vaccination with a novel Haemophilus influenzae-Neisseria meningitidis serogroup C conjugate vaccine. Clin Vaccine Immunol. 2007 Apr;14(4):426-34. doi: 10.1128/CVI.00377-06. Epub 2007 Feb 7. PMID 17287313
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 711202/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 711202/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 711202/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 711202/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 711202/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 711202/008 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register